CLINICAL TRIAL: NCT02565966
Title: Understanding the Mechanism(s) of Action on the Modified Atkins Diet for Epilepsy: Human Brain Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: St. Barnabas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-01069
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Modified Atkins Diet (MAD) (Experimental)
  Interventions: Other: Modified Atkins Diet (MAD)
- Normal Diet (No Intervention): Those patients in the normal diet (no intervention) group will also meet with the epilepsy center nutritionist to review the food diary and completion of this document, similar to those in the intervention (MAD) group. No dietary restrictions will be made in this group.

INTERVENTIONS:
Other: Modified Atkins Diet (MAD) — For those in the MAD intervention group, the dietitian trains the patient and family in the preparation and management of this specialized therapy including sick-day guidelines, meal planning, carbohydrate counting and trouble-shooting. Written and verbal education including, but not limited to: recipes, education materials, sample meal plans and carbohydrate counters are provided to the patient during the initial education session. The caregiver/patient is trained in the outpatient setting and the diet is implemented at home with as much email/phone support from the dietician and ketogenic team as the patient needs to successfully maintain the diet. Medications are all changed over to the lowest carbohydrate forms to eliminate excess carbohydrate intake and all patients are started on vitamin supplements to maintain adequate nutrition.
  Arms: Modified Atkins Diet (MAD)

SUMMARY:
The purpose of this study is to better define the potential molecular and anti-inflammatory changes induced by the modified Atkins diet in the brains of patients with treatment resistant epilepsy. The investigators plan to enroll 30 subjects overall in this study to compare serologic and brain tissue specimens. At NYU, investigators plan to enroll 20 subjects; an estimated ten (10) subjects will consume a modified Atkins diet for 3-4 weeks prior to surgery and an estimated ten (10) subjects will consume a non-modified, higher carbohydrate diet. Investigators at Saint Barnabas Medical Center plan to enroll 10 subjects in this study to compare serologic and brain tissue specimens. Approximately five (5) subjects will consume a modified Atkins diet for 3-4 weeks prior to surgery and five (5) subjects will consume a non-modified, higher carbohydrate diet. Blood and brain tissue specimens will be obtained at the time of surgery and will be compared. The goal of this study is to identify whether or not there are changes in neuroinflammation or neuroexcitability in the human brain induced by the modified Atkins diet.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for epilepsy surgery at New York Langone Medical Center or St Barnabas Medical Center will be eligible for enrollment.

* Patient is at least 18 years of age
* Patient is willing to participate by complying with the modified Atkins diet 3 - 4 weeks prior to surgery and maintain a thorough food diary (Intervention study group) or to continue their usual diet and maintain a thorough food diary (Nonintervention study group)
* Patient/ his/her parent, caregiver, or health care proxy is willing and able to provide consent or assent

Exclusion Criteria:

* Patients under the age of 18 will be excluded
* Patients in whom a two-stage surgery is planned without any resection of brain tissue during the initial craniotomy
* Patients unwilling to comply with modified Atkins diet 3 -4 weeks prior to surgery or unwilling to maintain a thorough food diary will be excluded.
* Patients who are currently on an Atkins or Low Glycemic Index Diet will not be eligible for inclusion in the nonintervention group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Neuroinflammation markers in blood | At time of surgery (approximately 3-4 weeks after randomization)
  As measured by level of cytokines IL-6, TNF alpha, and C-reactive protein in blood samples
Metabolism | At time of surgery (approximately 3-4 weeks after randomization)
  As measured by level of fasting lipid profile, acylcarnitine profile, and beta-hydroxybutyrate in blood
Neuroinflammation markers in brain tissue | At time of surgery (approximately 3-4 weeks after randomization)
  As measured by level of cytokines, IL6, TNF alpha, and microglial activation and proliferation in brain tissue obtained during durgery
Levels of leptin in brain tissue | At time of surgery (approximately 3-4 weeks after randomization)
Levels of adenosine in brain tissue | At time of surgery (approximately 3-4 weeks after randomization)
Levels of adenosine kinase in brain tissue | At time of surgery (approximately 3-4 weeks after randomization)
Levels of adenosite-1 (A1) receptors in brain tissue | At time of surgery (approximately 3-4 weeks after randomization)
Levels of enzymes that synthesize glutamate and GABA | At time of surgery (approximately 3-4 weeks after randomization)
  As measured in brain tissue obtained during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Orrin Devinsky, MD, Principal Investigator — NYU Langone Epilepsy Center
Locations (2):
- United States (2):
  - Institute of Neurology and Neurosurgery at Saint Barnabas, Livingston, New Jersey
  - NYU Langone Epilepsy Center, New York, New York

REFERENCES:
- [Derived] Leitner DF, Siu Y, Korman A, Lin Z, Kanshin E, Friedman D, Devore S, Ueberheide B, Tsirigos A, Jones DR, Wisniewski T, Devinsky O. Metabolomic, proteomic, and transcriptomic changes in adults with epilepsy on modified Atkins diet. Epilepsia. 2023 Apr;64(4):1046-1060. doi: 10.1111/epi.17540. Epub 2023 Feb 24. PMID 36775798